CLINICAL TRIAL: NCT02960347
Title: Examining the Efficacy of tDCS in the Attenuation of Epileptic Paroxysmal Discharges and Clinical Seizures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herzog Hospital (Other)
Collaborators: The City College of New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Meiron 2013-4
Record Dates: First submitted 2016-11-01; First posted 2016-11-09 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2016-11

CONDITIONS: Ohtahara Syndrome
MeSH Terms: conditions — Infantile Epileptic-Dyskinetic Encephalopathy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active tDCS (Experimental): open label active tDCS treatment
  Interventions: Device: High-definition (HD) transcranial direct current stimulator, HD-tDCS with 4x1 HD adaptor

INTERVENTIONS:
Device: High-definition (HD) transcranial direct current stimulator, HD-tDCS with 4x1 HD adaptor — Non-invasive focal neuromodulation
  Other Names: tDCS

SUMMARY:
The current study examined the feasibility of High-Definition tDCS (HD-tDCS) in reducing epileptiform activity in a 30-month-old child suffering from early onset epileptic encephalopathy. HD-tDCS was administered over 10 intervention days spanning two weeks including pre- and post-intervention video-electroencephalography (EEG) monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Initial diagnosis of Ohtahara syndrome/West syndrome/ Lennox-Gastaut syndrome by a pediatric neurologist using video-EEG
2. Ongoing synchronous Hypsarrhythmia
3. Modified Hypsarrhythmia with a consistent focus of paroxysmal discharges
4. Signed informed consent of parents/immediate legal guardian
5. Age 10 to 36 months
6. Infant should be in a steady state indicated by a baseline test of electrolytes and biochemistry blood test, heart rate, temperature, respiratory rate, and saturation.

Exclusion Criteria:

1. Metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
2. History of adverse reaction to neurostimulation
3. Significant ECG abnormality

Ages: 10 Months to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
change in seizure frequency from baseline | day 1, day 3, day 5, day 6, day 8, day 10, day 13, day 20, day 27, day 33, day 40, day 50

CONTACTS AND LOCATIONS:
Overall Officials: Rena Gale, MD, Principal Investigator — Herzog Hospital
Locations (1):
- Herzog Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Auvichayapat N, Sinsupan K, Tunkamnerdthai O, Auvichayapat P. Transcranial Direct Current Stimulation for Treatment of Childhood Pharmacoresistant Lennox-Gastaut Syndrome: A Pilot Study. Front Neurol. 2016 May 4;7:66. doi: 10.3389/fneur.2016.00066. eCollection 2016. PMID 27199889
- [Result] Sunderam S, Gluckman B, Reato D, Bikson M. Toward rational design of electrical stimulation strategies for epilepsy control. Epilepsy Behav. 2010 Jan;17(1):6-22. doi: 10.1016/j.yebeh.2009.10.017. Epub 2009 Nov 17. PMID 19926525
- [Result] Kessler SK, Minhas P, Woods AJ, Rosen A, Gorman C, Bikson M. Dosage considerations for transcranial direct current stimulation in children: a computational modeling study. PLoS One. 2013 Sep 27;8(9):e76112. doi: 10.1371/journal.pone.0076112. eCollection 2013. PMID 24086698
- [Result] Yook SW, Park SH, Seo JH, Kim SJ, Ko MH. Suppression of seizure by cathodal transcranial direct current stimulation in an epileptic patient - a case report -. Ann Rehabil Med. 2011 Aug;35(4):579-82. doi: 10.5535/arm.2011.35.4.579. Epub 2011 Aug 31. PMID 22506177
- [Result] Datta A, Bansal V, Diaz J, Patel J, Reato D, Bikson M. Gyri-precise head model of transcranial direct current stimulation: improved spatial focality using a ring electrode versus conventional rectangular pad. Brain Stimul. 2009 Oct;2(4):201-7, 207.e1. doi: 10.1016/j.brs.2009.03.005. PMID 20648973
- [Derived] Meiron O, Gale R, Namestnic J, Bennet-Back O, Gebodh N, Esmaeilpour Z, Mandzhiyev V, Bikson M. Antiepileptic Effects of a Novel Non-invasive Neuromodulation Treatment in a Subject With Early-Onset Epileptic Encephalopathy: Case Report With 20 Sessions of HD-tDCS Intervention. Front Neurosci. 2019 May 29;13:547. doi: 10.3389/fnins.2019.00547. eCollection 2019. PMID 31191235